CLINICAL TRIAL: NCT03041129
Title: Post-Prandial Liver Glucose Metabolism in Polycystic Ovarian Syndrome (PCOS) and Understanding Standard of Care Medications
Brief Title: Post-Prandial Liver Glucose Metabolism in PCOS
Acronym: PLUM
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2399
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Polycystic Ovarian Syndrome; Obesity; Hepatic Steatosis
Keywords: hepatic de novo lipogenesis
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Fatty Liver | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA for hepatic steatosis related genes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Untreated PCOS: PCOS per NIH criteria. Obese Lifestyle treatment only.
  Interventions: Diagnostic Test: oral glucose tolerance test; Diagnostic Test: MRI of liver
- Metformin PCOS-(Study arm not funded): PCOS per NIH criteria. Obese Taking 1500 mg of metformin or more per day for at least 6 months.
  Interventions: Diagnostic Test: oral glucose tolerance test; Diagnostic Test: MRI of liver
- Oral Contraceptive PCOS-(Study arm not funded): PCOS per NIH criteria. Obese Taking 30 mcg of ethanyl estradiol or more per day for at least 6 months.
  Interventions: Diagnostic Test: oral glucose tolerance test; Diagnostic Test: MRI of liver
- Obese Control group-(Study arm not funded): Obese Regular menses at least 18 months post-menarche Females only
  Interventions: Diagnostic Test: oral glucose tolerance test; Diagnostic Test: MRI of liver

INTERVENTIONS:
Diagnostic Test: oral glucose tolerance test — 6 hours OGTT
Diagnostic Test: MRI of liver — MRI of the liver and use of DIXON method

SUMMARY:
The Investigators will measure if hepatic metabolism is upregulated in obese girls with PCOS and hepatic steatosis (HS), compared to PCOS without HS and obese controls without HS.

DETAILED DESCRIPTION:
This will be a cross-sectional study with 4 groups of youth. A 6 hour OSTT (Oral Sugar Tolerance Test) with an oral U-C13 glycerol tracer will be paired with nuclear magnetic resonance spectroscopy (NMR) isotopomer analysis of serum samples to describe flux through the hepatic pentose phosphate pathway, TCA cycle and FAS pathways in girls with PCOS receiving lifestyle only, metformin or oral contraceptive treatment, and obese girls with regular menses receiving lifestyle therapy. Hepatic steatosis will be measured with MRI.

Please note that 3 study groups: PCOS on metformin, PCOS on oral contraceptive treatment, and obese girls with regular menses were not funded in the study, so no participants were enrolled in these 3 arms of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Ages 12-21
3. Sedentary- less than 2.5 hours of moderate (jogging, swimming etc) exercise a week.
4. BMI equal or greater than the 90th percentile for age and gender
5. For PCOS groups:

   * (NIH definition) irregular menstrual cycles at least 1.5 years after menarche, and
   * either clinical evidence of hyperandogenism, or
   * elevated Testosterone (above the norms for age/tanner stage) at time of screening, or documented prior to initiation of therapy for OCP and metformin groups.
6. For PCOS groups:

   * patients un-treated or currently treated with either Metformin 1500-2000 mg a day, or
   * oral contraception (30-35 mcg ethynyl estradiol a day) for at least 6 months, with > 80% adherence confirmed via refill frequency from pharmacy.
7. For non-PCOS groups:

   * regular menstrual cycles at least 1.5 years after menarche, and
   * no clinical evidence of hyperandrogenism.

Exclusion Criteria:

1. Use of medications known to affect insulin sensitivity:

   * oral glucocorticoids within 10 days,
   * atypical antipsychotics,
   * immunosuppressant agents,
   * HIV medications.
   * Nexplanon, Depo-Provera or Mirena progesterone only contraceptives.
   * Dermal patch or vaginal ring contraception methods.
   * For controls only: metformin or oral contraception.
2. Currently pregnant or breastfeeding women. Development of pregnancy during the study period will necessitate withdrawal from the study.
3. Severe illness requiring hospitalization within 60 days
4. Diabetes, defined as Hemoglobin A1C > 6.4%
5. BMI percentile less than the 90th percentile for age and sex.
6. Weight >325 lbs or <84 lbs.
7. Anemia, defined as Hemoglobin < 10 mg/dL
8. Diagnosed major psychiatric or developmental disorder limiting informed consent
9. Implanted metal devices that are not compatible with MRI
10. Use of blood pressure medications
11. Known liver disease other than NAFLD or AST or ALT >150 mg/mL

    -

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Females only
Study Population: Girls age 12-21. Obese >90th percentile for BMI for age.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Cree-Green, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anshutz Medical Campus/Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carreau AM, Pyle L, Garcia-Reyes Y, Rahat H, Vigers T, Jensen T, Scherzinger A, Nadeau KJ, Cree-Green M. Clinical prediction score of nonalcoholic fatty liver disease in adolescent girls with polycystic ovary syndrome (PCOS-HS index). Clin Endocrinol (Oxf). 2019 Oct;91(4):544-552. doi: 10.1111/cen.14062. Epub 2019 Aug 16. PMID 31301251

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Untreated PCOS | Metformin PCOS-(Study Arm Not Funded) | Oral Contraceptive PCOS-(Study Arm Not Funded) | Obese Control Group-(Study Arm Not Funded)
Started | 19 | 0 | 0 | 0
Completed | 17 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only participants enrolled in the untreated PCOS group. No participants were enrolled in the other arms of the study due to funding.
Groups:
- Total: Total of all reporting groups
Arm/Group | Untreated PCOS | Metformin PCOS-(Study Arm Not Funded) | Oral Contraceptive PCOS-(Study Arm Not Funded) | Obese Control Group-(Study Arm Not Funded) | Total
Number analyzed (Participants) | 17 | 0 | 0 | 0 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.2 (1.68) |  |  |  | 16.2 (1.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 |  |  |  | 17
  Male | 0 |  |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 0 | 0 | 0 | 10
  Not Hispanic or Latino | 7 | 0 | 0 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 |  |  |  | 17

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Fat Fraction
Description: Amount of fat in the liver measured by MRI and calculated via the Dixon method as the proton density hepatic fat fraction, which ranges from 0-75%. Greater than 5% is considered extra fat in the liver.
Time Frame: Measured up to 4 months from enrollment
Population: Adolescent females with dx of PCOS
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Untreated PCOS | Metformin PCOS-(Study Arm Not Funded) | Oral Contraceptive PCOS-(Study Arm Not Funded) | Obese Control Group-(Study Arm Not Funded)
Number analyzed (Participants) | 17 | 0 | 0 | 0
Percent | 8.35 (7.55) |  |  |

2. Secondary Outcome: Hepatic Metabolism Ratios
Description: Percent indirect glucose at 360 minutes following an oral sugar tolerance test (OGTT) with an isotope labeled oral glycerol tracer.
Time Frame: Measured up to 4 months from enrollment
Population: Adolescent females with diagnosis of PCOS
Measure: Mean (Standard Deviation); unit: percentage of indirect glucose
Arm/Group | Untreated PCOS | Metformin PCOS-(Study Arm Not Funded) | Oral Contraceptive PCOS-(Study Arm Not Funded) | Obese Control Group-(Study Arm Not Funded)
Number analyzed (Participants) | 16 | 0 | 0 | 0
percentage of indirect glucose | 22.1 (6.9) |  |  |

3. Secondary Outcome: Whole Body Insulin Sensitivity
Description: Participants will undergo a 75 gram oral glucose tolerance test, and whole body insulin sensitivity will be expressed as Si, calculated via the oral minimal model.
Time Frame: Measured up to 4 months from enrollment
Population: Adolescent females with dx of PCOS
Measure: Mean (Standard Deviation); unit: dL/kg/min per uU/mL
Arm/Group | Untreated PCOS | Metformin PCOS-(Study Arm Not Funded) | Oral Contraceptive PCOS-(Study Arm Not Funded) | Obese Control Group-(Study Arm Not Funded)
Number analyzed (Participants) | 17 | 0 | 0 | 0
dL/kg/min per uU/mL | 0.000278106 (0.000393419) |  |  |

4. Secondary Outcome: Sleep Duration
Description: Sleep duration will be assessed using home actigraphy using the Philips Actigraph wrist-worn watch, and collects 7 days of data.
Time Frame: Measured up to 4 months from enrollment
Population: Adolescent females with dx of PCOS
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Untreated PCOS | Metformin PCOS-(Study Arm Not Funded) | Oral Contraceptive PCOS-(Study Arm Not Funded) | Obese Control Group-(Study Arm Not Funded)
Number analyzed (Participants) | 14 | 0 | 0 | 0
Minutes | 443.44 (52.63) |  |  |

5. Secondary Outcome: Sleep Quality
Description: Apnea Hypopnea Index (AHI) will be measured using WatchPAT. The higher the AHI, indicates more severe sleep apnea.
  The AHI is the number of times you have apnea or hypopnea during one night, divided by the hours of sleep.
  Normal sleep: An AHI of fewer than five events, on average, per hour Mild sleep apnea: An AHI of five to 14 events per hour Moderate sleep apnea: An AHI of 15 to 29 events per hour Severe sleep apnea: An AHI of 30 or more events per hour
Time Frame: Measured up to 4 months from enrollment
Population: Adolescent females with dx of PCOS
Measure: Mean (Standard Deviation); unit: Apnea Hypoxia Index
Arm/Group | Untreated PCOS | Metformin PCOS-(Study Arm Not Funded) | Oral Contraceptive PCOS-(Study Arm Not Funded) | Obese Control Group-(Study Arm Not Funded)
Number analyzed (Participants) | 17 | 0 | 0 | 0
Apnea Hypoxia Index | 19.66 (10.82) |  |  |

6. Secondary Outcome: Hepatic Phosphate Concentrations
Description: 31 phosphorus spectroscopy will be utilized to measure hepatic Phosphodiesterase (PDE)/Total phosphate concentration. This is measured in the MRI using a phosphorus coil.
Time Frame: Measured up to 4 months from enrollment
Population: Untreated PCOS, All participants whom the scan worked for. Did not work in those with a large waist circumference
Measure: Mean (Standard Deviation); unit: percentage of PDE/total phosphate
Arm/Group | Untreated PCOS | Metformin PCOS-(Study Arm Not Funded) | Oral Contraceptive PCOS-(Study Arm Not Funded) | Obese Control Group-(Study Arm Not Funded)
Number analyzed (Participants) | 15 | 0 | 0 | 0
percentage of PDE/total phosphate | 23 (7) |  |  |

ADVERSE EVENTS:
Time Frame: 9 days. Participants wore a couple of watches at home for 7 days and the metabolic study was 2 days long.
Description: Adverse events only reported for the untreated PCOS group, since no participants were enrolled in the other groups.
Arm/Group | Untreated PCOS | Metformin PCOS-(Study Arm Not Funded) | Oral Contraceptive PCOS-(Study Arm Not Funded) | Obese Control Group-(Study Arm Not Funded)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/17 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to the Covid-19 outbreak, and lack of funding we were unable to enroll the participants in the metformin arm, oral contraceptive arm, and the obese control group. Only enrolled participants in untreated PCOS group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03041129/Prot_SAP_000.pdf